CLINICAL TRIAL: NCT06529172
Title: Effects of Resistance Training, Yijinjing and Baduanjin Exercise on Bone Mineral Density and Bone Metabolism in Older Women
Brief Title: Bone Mineral Density and Bone Metabolism in Older Women
Acronym: BMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng Liang (Other)
Collaborators: Chengdu Sport University (Other)
Responsible Party: Sponsor-Investigator, Cheng Liang, Pro, Chengdu Sport University
Organization: Chengdu Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ChengduSU; Youth Found of Humanities and (Other: Education of China)
Record Dates: First submitted 2024-07-25; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis, Age-Related
Keywords: bone mineral density; bone metabolism
MeSH Terms: conditions — Osteoporosis | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): The CG group maintained their original lifestyle without engaging in regular exercise.
  Interventions: Other: Resistance training; Other: Yijinjing; Other: Baduanjing; Other: Control
- Resistance training (Experimental): RT group (RG, n = 21), YJJ group (YG, n = 22), BDJ group (BG, n = 21). These groups performed the assigned exercises for 24 weeks (3 times/week, 60 min/time).
  Interventions: Other: Resistance training; Other: Yijinjing; Other: Baduanjing; Other: Control
- Yijinjing (Experimental): RT group (RG, n = 21), YJJ group (YG, n = 22), BDJ group (BG, n = 21). These groups performed the assigned exercises for 24 weeks (3 times/week, 60 min/time).
  Interventions: Other: Resistance training; Other: Yijinjing; Other: Baduanjing; Other: Control
- Baduanjing (Experimental): RT group (RG, n = 21), YJJ group (YG, n = 22), BDJ group (BG, n = 21). These groups performed the assigned exercises for 24 weeks (3 times/week, 60 min/time).
  Interventions: Other: Resistance training; Other: Yijinjing; Other: Baduanjing; Other: Control

INTERVENTIONS:
Other: Resistance training — RG performed RT with an elastic band (yellow, force of 9-11 pounds when stretched twice the original length). They performed eight movements. Each movement was performed for 3-5 sets at 8 times/sets with 30 s of rest between groups. The movements included upright rows, reverse curls, standing shoulder rotations, neck-elbow extensions, elbow bends, downward lunges, standing leg lifts, side lifts and standing back kicks. All participants completed the RT movements according to the regular rhythm (1-2-1) provided by the experimenter, which ensured that all participants had similar movements completion rates.
Other: Yijinjing — YG performed 12 movements . These movements included extending the hands upwards and slowly lowering them; extending the torso by stretching the hands straight up and bending the body to the left or right; squatting with the hands on the knees and standing up slowly; bending the body to the left or right side, extending the arms and waist; getting down on the knees, leaning forward, extending the hands forward and slowly pulling them back; bending forward, placing the hands around the knees and standing up slowly; placing the hands on the hips; and leaning back to stretch the back and waist.
Other: Baduanjing — BG performed eight movements . These movements included holding the hands straight up, slowly bringing the hands down and turning the waist while in a standing position; bending the body to the left or right side and extending the arms; extending one hand straight up, placing the other hand on the waist, then switching arms and repeating the movement; tilting the head back and looking back while stretching the neck and back; squatting the body, swinging the head and hips from side to side and moving the spine and waist; bending the body forward, touching the hands to the toes and standing up slowly; making fists with the hands and moving the arms and shoulders; and gently bouncing the body to relax the whole body in a standing position.
Other: Control — The CG group maintained their original lifestyle without engaging in regular exercise

SUMMARY:
The objective of this study is to assess the impact of different exercise interventions on bone mineral density (BMD) in older women. It will also evaluate the safety and compliance of these interventions. The primary questions it aims to address are:

Does resistance training, Yijinjing, or Baduanjin improve BMD in postmenopausal women? What are the compliance rates and any adverse effects associated with these exercise programs? Participants will be divided into 4 groups and compared against a control group that maintains their usual lifestyle.

Participants will:

Engage in their assigned exercise program three times a week for 24 weeks Receive calcium and vitamin D supplementation daily Keep a log of exercise adherence and any side effects experienced The study will utilize the International Physical Activity Questionnaire and dual-energy X-ray absorptiometry for comprehensive assessments.

DETAILED DESCRIPTION:
The calculation revealed that a minimum number of 80 participants was required. In this study, the investigators employed a straightforward randomization method for group allocation. This study designated four sets of cards numbered 1 to 4, with each number representing one of the groups: RT group (RG), YJJ group (YG), BDJ group (BG) and control group (CG). Each set included 23 cards, and participants were assigned to groups using a draw from these sets, ensuring random and equal distribution across groups.

Participants were required to engage in exercise sessions conducted in a centralized manner, with three 60-minute sessions per week. The investigators did indeed monitor and document the compliance of the participants. Compliance encompassed adherence to the exercise regimen, intake of supplements, and compliance with all other research requirements. The majority of participants demonstrated good compliance throughout the 24-week study period.

Exercise intervention The initial exercise intervention was provided as follows: throughout the entire intervention period, the four groups of participants were administered calcium and vitamin D supplementation (produced by Wyeth Pharmaceuticals; specification: 600 mg per tablet; National Medicine Permission No. H10950029, once in the morning and once in the evening, one tablet each time). During the intervention period, participants were advised to avoid smoking and the consumption of alcohol, coffee, strong tea, and carbonated drinks. The CG group maintained their original lifestyle without engaging in regular exercise. The intervention period lasted for 24 weeks with a frequency of three times per week. Each session lasted for 60 min and included approximately 10 min of preparatory activities, warm-up and relaxation. Exercise intensity was based on the research method by Cheng et al. with the heart rate controlled at (220 - age) × (55% to 70%). After each exercise session, the carotid pulse was recorded by manually counting the beats over a 30-second period post-exercise, using this data to adjust the exercise intensity if it deviated from the target heart rate range.

RG performed RT with an elastic band (yellow, force of 9-11 pounds when stretched twice the original length). They performed eight movements. Each movement was performed for 3-5 sets at 8 times/sets with 30 s of rest between groups. The movements included upright rows, reverse curls, standing shoulder rotations, neck-elbow extensions, elbow bends, downward lunges, standing leg lifts, side lifts and standing back kicks. All participants completed the RT movements according to the regular rhythm (1-2-1) provided by the experimenter, which ensured that all participants had similar movements completion rates.

YG performed 12 movements. These movements included extending the hands upwards and slowly lowering them; extending the torso by stretching the hands straight up and bending the body to the left or right; squatting with the hands on the knees and standing up slowly; bending the body to the left or right side, extending the arms and waist; getting down on the knees, leaning forward, extending the hands forward and slowly pulling them back; bending forward, placing the hands around the knees and standing up slowly; placing the hands on the hips; and leaning back to stretch the back and waist.

BG performed eight movements. These movements included holding the hands straight up, slowly bringing the hands down and turning the waist while in a standing position; bending the body to the left or right side and extending the arms; extending one hand straight up, placing the other hand on the waist, then switching arms and repeating the movement; tilting the head back and looking back while stretching the neck and back; squatting the body, swinging the head and hips from side to side and moving the spine and waist; bending the body forward, touching the hands to the toes and standing up slowly; making fists with the hands and moving the arms and shoulders; and gently bouncing the body to relax the whole body in a standing position.

The first 4 weeks of YG and BG were the learning period, and weeks 5-24 weeks were the consolidation and strengthening period. During the consolidation and strengthening period, the participants were required to practise six sets of movements each time with a gap of approximately 30 s. With the increase in intervention weeks, the participants can appropriately adjust the stretching length of the elastic band and increase the number of sets to control the load in accordance with their own condition. The experimenter conducted weekly interviews, in person or via telephone, using a standardized questionnaire to document all participants' living conditions. The recorded information mainly involved the participants' eating habits (diet variety and amount), working and resting patterns (sleep quality, sunshine amount and residence area) , whether the participants took other regular exercise and whether the participants took drugs that affected BMD. Diet and Lifestyle Interview Findings: This study found that participants largely adhered to their regular dietary habits and physical activity levels throughout the study. This consistency suggests that these factors were not significant confounders affecting the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Females who were aged 60-70 years
* Recently expressed willingness to engage in fitness activities
* Passed a health examination
* Signed an informed consent form in accordance with the Helsinki Declaration were included.

Exclusion Criteria:

* Heart disease
* History of severe lower limb injury
* A T-score of less than -2.5 standard deviations is diagnostic of osteoporosis
* Currently taking antiosteoporosis medication
* Currently taking hormone replacement therapy
* Engaging in other regular forms of exercise were excluded.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry measurements | 24 Weeks
  A Norland XR-46 dual-energy X-ray BMD tester was used to measure the BMD of the lumbar L2-4 and proximal femur of the dominant side (femur neck, greater trochanter and Ward's triangle). Five non-re-entrant scans were performed at each measurement site. The error coefficients of the measurement location were 1-2% in the lumbar L2-4, femoral neck and greater trochanter and 2.5-5% in Ward's triangle. The coefficient of variation in the lumbar vertebrae and the proximal femur was 1.1% and 1.85%, respectively.
Serum bone metabolism markers | 24 Weeks
  Fasting venous blood (5 ml) was drawn between 7 a.m. and 8 a.m. at both baseline and after 24 weeks, with samples subsequently centrifuged at 3000 r/min for 5 minutes in each instance. Serum levels of PINP, OC, and β-CTX were measured using an automatic chemiluminescence analyzer, the LIAISON® XL, which is manufactured by the Italian company DiaSorin. The kit required for the experiment was purchased from Nanjing Jiancheng Bioengineering Institute and utilised in strict accordance with its instructions.

SECONDARY OUTCOMES:
Physical Activity Assessment | 24 Weeks
  This study incorporated a validated assessment tool to monitor the participants' physical activity levels. For all groups, we utilized the International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Liang Cheng, Dr, Study Director — Chengdu Sport University
Locations (1):
- Chengdu Sport University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No